CLINICAL TRIAL: NCT03007433
Title: Assessment of Gastric Motor and Sensory Function to a Large Test Meal by Gamma Scintigraphy, Magnetic Resonance Imaging and a Nutrient Drink Test in Health and Patients With Functional Dyspepsia
Brief Title: Assessment of GI Function to a Large Test Meal by Non-invasive Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10GA007; 10/H0408/52 (Other: Research ethics committee)
Record Dates: First submitted 2016-11-21; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Functional Dyspepsia
Keywords: gastric emptying; functional dyspepsia; non invasive imaging; MRI; gamma scintigraphy; gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy volunteers (Experimental): 60 healthy volunteers with no functional dyspepsia as defined by the Rome Questionnaire and no more than mild symptoms on maximum 1 days a week on the GSRS, that meet inclusion and exclusion criteria will be recruited. Eligible subjects will be block randomized by sex and age such that 10 men and women in each age group (<40, 41-60, >60) are recruited.
  Interventions: Other: 400ml of Liquid Nutrient Drink
- Functional dyspeptic patients (Experimental): 20 patients with functional dyspepsia with postprandial distress syndrome as defined by the Rome IV Questionnaire and at least moderate symptom severity on at least 3 days a week that meet the inclusion and exclusion criteria will be recruited to provide pilot data in the local patient population
  Interventions: Other: 400ml of Liquid Nutrient Drink

INTERVENTIONS:
Other: 400ml of Liquid Nutrient Drink — 12MBq Technetium-99m-DTPA will be added as a non-absorbable marker incorporated into liquid nutrient drink Fortisip Vanilla (Nutricia Clinical)
  Other Names: Fortisip Vanilla

SUMMARY:
Dyspeptic symptoms such as abdominal pain, bloating and nausea after a meal are common; however the cause of these problems in many patients is often unclear despite medical investigation. This is because "dyspeptic symptoms" are only rarely related to acid reflux, stomach ulcers or cancer that can be diagnosed by endoscopy. Rather, the cause is abnormal stomach function, so-called "functional dyspepsia", a condition in which the digestive system does not function normally after a meal. Gastric scintigraphy is the standard investigation of stomach function in patients with this condition. It involves eating a small test meal that includes a tiny dose of radioactive material so that the movement of food can be visualised as it empties from the stomach. An important limitation of this approach is that symptoms are rarely caused and delayed emptying after a small meal is present only in a minority of patients and, thus, the ability of this investigation to explain the cause of symptoms or guide medical treatment is limited.

This research project is designed to compare three new investigations of stomach function using a relatively large meal. This information will help to explain the causes of symptoms after a meal. The investigations to be tested include: (1) Nutrient Drink Test, (2) Gastric Scintigraphy and (3) Magnetic Resonance Imaging. All three tests are safe, easy to perform and non-invasive (i.e. do not involve inserting catheters through the nose and into the stomach or taking blood). The results should provide more useful information to doctors looking after patients with dyspeptic symptoms.

This study will compare test results from healthy volunteers, with patients attending clinic for investigation of dyspeptic symptoms. The aim is to document abnormal function of the stomach and intestines and to identify the causes of dyspeptic symptoms after a meal.

DETAILED DESCRIPTION:
The Nutrient Drinking Test will be performed as part of the screening visit to ensure that all patients that consent to participate in the full study are able to complete the imaging studies that require ingestion of 400ml liquid nutrient (Fortisip Vanilla (Nutricia Clinical) diluted 1:1 with water to 0.75kcal/ml, 4.5g fat/100ml).

Subjects will drink one from a series of beakers containing 40ml liquid nutrient every minute. During the drinking test, subjects will score satiety, fullness, bloating, heartburn, nausea and epigastric pain at 5-min intervals using a 100mm visual analogue scale (sample attached). Participants will be instructed to cease intake when they reported maximal satiety or very severe dyspeptic symptoms (defined as VAS score of >90 mm). The total volume ingested will be recorded. Symptoms will be assessed again 15 and 30 min after cessation of intake.

If the subject fulfils the inclusion and exclusion criteria including ingestion of ≥400ml at the drinking test and consents to continue then appointments will be made for gamma scintigraphy and MRI studies according to a prospective randomization plan.

MRI Study Day After eligibility has been confirmed subjects will ingest the paramagnetic contrast labelled liquid nutrient test meal according to a standardized protocol. Subjects will drink one from a series of ten beakers containing 40ml liquid nutrient every minute. During the test meal, subjects will score satiety, fullness, bloating, heartburn, nausea and epigastric pain at baseline, 5 and 10 minute using a visual analogue scale (VAS 0-100 mm). These measurements will be repeated at 30min and at the conclusion of the imaging study (see below).

Studies will be performed using a 1.5T whole MRI system (Intera, Philips, Best, The Netherlands). Six rectangular surface coils (height = 20 cm, width = 10 cm), fixed around the abdomen and connected to independent receive channels were used for signal detection.

Gamma Scintigraphy Study Day After eligibility has been confirmed subjects will ingest the radiolabelled liquid nutrient test meal according to a standardized protocol. Subjects will drink one from a series of ten beakers containing 40ml liquid nutrient every minute. During the test meal, subjects will score satiety, fullness, bloating, heartburn, nausea and epigastric pain at baseline, 5 and 10 min using a visual analogue scale (VAS 0-100 mm).

ELIGIBILITY:
Inclusion Criteria:

* Be an adult patient above 18 years old
* Meet the block randomization criteria for age and sex (no such allocation required for patient group)
* Have a body mass index of >18 and <30kg.m2 and not exceed a waist circumference of 99cm at 5cm above ileal crest
* Be able to give voluntary informed consent and from whom written consent to participate has been obtained.
* Be able to understand the study, willing to co-operate with the study procedures and able to attend all study assessments.
* Be willing to abstain from alcohol for 24 hours before and during the imaging appointment.
* Be willing to fast from midnight prior to the screening and imaging appointment
* Be able to ingest at least 400ml nutrient liquid (0.75kcal/ml at 40ml/min) during a Nutrient Drinking Test without experiencing more than moderate dyspeptic symptoms (no such restriction for patients with dyspeptic symptoms)
* Be willing to consent to their General Practitioner (GP) being informed of their participation.

Exclusion Criteria:

* Have a history of gastrointestinal disease or surgery (other than appendicitis or hysterectomy)
* Have ongoing disease requiring active management
* Have a documented history of alcohol or drug abuse
* Fail to satisfy the investigator's assessment of fitness to participate based on a survey of inclusion and exclusion criteria
* Have consumed alcohol within 24 hours of start of study
* Have participated in a similar study involving the use of radioisotopes in the previous 3 months such that participating in the current study would exceed the recommended yearly exposure limit (5mSv)
* Take any medication which may affect oesophageal or gastric motility for a minimum 7 days
* Have had previous history of gastric surgery
* Have active upper gastrointestinal diseases
* Have an active Eating Disorder
* Have an allergy to milk protein (milk based, lactose free test meal)
* Be a vegan
* Be pregnant or breastfeeding
* Have any contraindication to MRI scanning according to local guidelines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assessment of gastric sensory function using the nutrient drink test for volume ingested at maximum satiation | 4 months from consent
Estimate steady state gastric emptying rate (ml/min) using Gamma Scintigraphy And Magnetic Resonance Imaging (MRI) | 4 months from consent

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Fox, MD, Principal Investigator — Univeristy Hopsitals Nottingham
Locations (1):
- Nottingham University Hopsitals, Nottingham, Nottinghamshire, United Kingdom